CLINICAL TRIAL: NCT03984253
Title: Swiss Severe Asthma Register
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Jörg Leuppi (Other)
Collaborators: AstraZeneca (Industry); GlaxoSmithKline (Industry); Lungenliga Schweiz (Unknown); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Jörg Leuppi, Professor of Internal Medicine, Cantonal Hosptal, Baselland
Organization: Cantonal Hosptal, Baselland (Other)
Other Study IDs: 2018-01553
Record Dates: First submitted 2019-04-29; First posted 2019-06-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Severe Asthma
Keywords: Asthma; Severe; Register
MeSH Terms: conditions — Asthma; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Severe Asthma: All patients with severe asthma who will be treated in the participating centers should be continuously enrolled in the register.

SUMMARY:
Asthma is one of the most common chronic diseases. Asthma is characterized by chronic airway inflammation and associated with airway hyperresponsiveness and reversible airflow obstruction. The variability of airway obstruction is triggered by different factors that lead to a variety of different asthma phenotypes and subtypes. The various classification options for asthma (e.g. severity, by the predominantly existing inflammation or according to triggers), reflect its heterogeneity.

Despite improved therapeutic methods, the prevalence and morbidity of asthma has increased worldwide in the last years. Asthma is a serious and growing global health problem with around 300 million people affected, independent of age or sex. Estimated 250'000 people die prematurely each year due to their asthma.

Based on the SAPALDIA-study, the prevalence of Asthma in Switzerland is approximately 2-8%. Asthma is considered as a major factor in healthcare cost with up to CHF 1.2 billion per year. Asthma is not only a financial burden to a system; it affects the individual Quality of life negatively. Often health care professionals and patients underestimate the severity of the disease and overestimate asthma control. Severe asthma should not be equated with uncontrolled asthma. To reach a satisfying asthma control numerous factors need to be taken into consideration. Severe asthma is often associated with a high risk of frequent, severe exacerbations, which can even lead to death.

Several severe asthma cohorts and registries already exists and are reported in the literature. The aim of such registries is in general data collection and a better understanding of the disease. So far, most epidemiological studies on severe asthma are cross-sectional with no follow up measures. Only a few studies did repeated measures using the same methods.

Approximately 5% of all Asthma Patients suffers from severe asthma. These patients require systematic assessment and specialist care in dedicated respiratory centres. These centres have a key role in improving the outcome for severe asthma patients. At the same time they act as gatekeepers to ensure appropriate access to new, expensive therapies, this includes antibody treatment and interventional methods such as thermoplasty. These treatments require careful monitoring. It is important to ensure that they are given to the right population. Special assessment to monitor the efficacy and to prevent inappropriate prescribing, exposure of patients to unnecessary risks and excessive costs is indicated.

For all the mentioned reasons a Swiss Severe Asthma Register and a collaboration with an already existing register is needed to prospectively collect data about severe asthma in Switzerland.

DETAILED DESCRIPTION:
The overall objective is to establish a clinical register for patients with severe asthma. Since the number of patients with severe asthma at a single center is usually low, it will be important to collect data in a multi-center system to optimize the diagnostic evaluation and treatment of patients with severe asthma. So far, there is little reliable information about the frequency, phenotype and therapy of patients with severe asthma. The construction of a clinical register should close this gap. The primary objective is to show changes in symptoms control during follow up period and at study end by using the Asthma Control Test (ACT). Secondary endpoints are to collect data to better understand asthma's natural history in patients with severe asthma. The examination will be based on the assessment of the parameters specified under "outcomes".

Patients presenting to participating study center (pulmonologists in private practice or in pulmonary departments in hospital within Switzerland) with severe asthma will be asked to take part in this study when corresponding to the eligibility criteria. All patients with severe asthma will be included in the register only after detailed information and written consent. After four months (for specific therapies) and after 12 months, patients should be re-evaluated for up to 15 years. These follow-up data will also be recorded in the register. During the follow-up visits, the same parameters will be collected as during the initial Baselineexamination (some parameters will be omitted, for example, therapy received or requested for the defined period of the last 12 months, etc.). Severe asthma patients receiving a new specific therapy, e.g. obtained with antibodies, but who cannot be included in the register with the complete parameter profile due to time or capacity reasons of the centers, should be recorded at least with defined basic data and a reduced number of parameters in the register. These parameters include according to the specific asthma approved specific therapies, socio-demographic data, lung function values, laboratory values, parameters of asthma control, smoking status and add-on- therapy. This should make it possible to record a subgroup of severe asthmatics that are suitable for antibody therapy and at the same time offer the attending physician the opportunity to adequately document these complex and expensive therapies by recording the defined parameters. In these patients, an evaluation of the therapy response should be carried out after four months and documented in the register. Thereafter, there is an annual follow-up. At any time, these patients can be transferred to the full version of the register by entering the missing parameters. Patients for whom only the basic data is available (basic version) as well as patients with complete parameter profile in the register are kept in the same database and can be evaluated together. In general, no register-specific examinations will be carried out, but only parameters anyway recorded routinely.

Since this is a cohort study, no sample size calculation can be calculated. Evaluations are carried out continuously. The collective of the data should be described by descriptive statistics concerning the basic data as well as the data of the function diagnostics. Subentities of severe asthma should be identified by a cluster analysis.

ELIGIBILITY:
Inclusion Criteria:

* In- and outpatients
* Age ≥ 0 year
* Informed consent as documented by signature

Adults:

"Asthma which requires treatment with guidelines suggested medications for GINA steps 4-5 asthma:

* High level therapy:

  1. high dose ICS with ≥ 1000 μg beclomethasone (powder) or equivalent in combination with LABA or leukotriene modifier/theophylline) for the previous year or
  2. Daily long-term therapy with systemic corticosteroids (CS) for ≥50% of the previous year to prevent it from becoming "uncontrolled" or which remains "uncontrolled" despite this therapy or
  3. Therapy with monoclonal antibodies independent from the co-therapy
* Middle level therapy:

Protokollsynopsis SAR Version 01 16.01.2019 Seite 4/10 a) Daily long-term therapy with medium-to high-dose ICS (≥500 μg Beclomethason (powder) or equivalent in combination with LABA or leukotriene modifier/theophylline) for the previous year and uncontrolled asthma defined as at least one of the following:

* Poor symptom control: ACQ consistently >1.5, ACT <20 (or "not well controlled" by NAEPP/GINA guidelines).
* Frequent severe exacerbations: two or more bursts of systemic CS (>3 days each) in the previous year.
* Serious exacerbations: at least one hospitalization, ICU stay or mechanical ventilation in the previous year.
* Airflow limitation: after appropriate bronchodilator withhold FEV1 <80% predicted (in the face of reduced FEV1/FVC defined as less than the lower limit of normal).
* Controlled asthma that worsens on tapering of these high doses of ICS or systemic CS (or additional biologics). The presence of any one of the following exclusion criteria will lead to exclusion of the patients:
* Life-expectancy <6 months
* Insufficient knowledge of project language

Children:

The criteria for severe or difficult asthma in children and adolescents are considered fulfilled in the case of insufficient symptom control in the last year despite medium/high antiinflammatory long-term therapy:

* age 0-18 years, at time of inclusion
* diagnosis of bronchial asthma made by a physician
* differential diagnoses excluded
* good compliance and trained inhalation technique
* treatment with biological approved for the treatment of severe asthma (currently only omalizumab) or

Proof of:

a) Positive Bronchodilation-test (≥12% increase in FEV1 after SABA) or b) Significant bronchial hyperresponsiveness after nonspecific provocation (e.g., with Methacholine or treadmill) according to ATS criteria (AJRCCM 2000)

* High level of therapy:

  1. Prolonged therapy with high dose inhaled steroid (ICS) (> 400 μg Budesonide equivalent /> 200 μg fluticasone alone); or
  2. Daily long-term therapy with medium- to high-dose ICS (≥ 400 μg Budesonide equivalent / ≥200 μg fluticasone) in combination with long-acting betaagonists and / or leukotriene receptor antagonist and / or theophylline; or
  3. Therapy with oral steroids fixed ≥3 last months.
* Insufficient asthma control

  a) Inadequate symptom control after NVL in the last 4 weeks: Protokollsynopsis SAR Version 01 16.01.2019 Seite 5/10
  * ≥3 x weekly asthma symptoms or use of ondemand medication; Or:
  * limited activity due to asthma; Or:
  * any symptoms at night; or b. Exacerbation(s) ≥1 last year that required treatment with systemic steroids and / or inpatient treatment c. limited lung function:
  * pathological Tiffeneau quotient or FEV1 at inclusion.
* Submission of a written consent (parent/ legal guardian).

Exclusion Criteria:

* Life-expectancy <6 months · Insufficient knowledge of project language

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to participating study center (pulmonologists in private practice or in pulmonary departments in hospital within Switzerland)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2034-02-28 (Estimated); Study Completion 2034-02-28 (Estimated)

PRIMARY OUTCOMES:
Symptom Control | Baseline, four months, yearly for up to 15 years
  Changes in symptom control at baseline and during the follow-up period and at study end using the Asthma Control Test (ACT).

SECONDARY OUTCOMES:
Exacerbations | Baseline, four months, yearly for up to 15 years
  Number of exacerbation with/without hospitalization
Utilization of the health care system | Baseline, four months, yearly for up to 15 years
  Number of Visits at one's general practitioner (GP) Number of Visits at a pneumologist/ specialist Number of emergency consultations Number of hospitalizations Number of rehabilitation stays
Quality of Life Questionnaire | Baseline, four months, yearly for up to 15 years
  Mini Asthma Quality of Life Questionnaire(Mini-AQLQ)
  * 15 Questions, Scale 1 to 7 , Minimum Score 15, Maximum Score 105.
  * The higher the Score is, the better the quality of life
Symptoms and health-related quality of life | Baseline, four months, yearly for up to 15 years
  Asthma Control Test 5 Questions, Scale 1- 5, Minimum score 5, max 25, the smaller the score the better is the Asthma control
Changes in Medication | Baseline, four months, yearly for up to 15 years
  Changes in Medication will be monitored for each subject. Changes in dose in mg Changes in substances if there is a new drug used.
Forced Vital Capacity (FVC) | Baseline, after four months, and after 12 months, then every year up to 15 years
  Changes in FVC in liter and % from the target value
Forced Exahled Volume in 1 second (FEV1) | Baseline, after four months, and after 12 months, then every year up to 15 years
  Changes in FEV1 in liter and % from the target value
Tiffeneau Test | Baseline, after four months, and after 12 months, then every year up to 15 years
  Changes in Tiffeneau in % and % from Target Value
Fraction of exhaled nitric oxide, FENO | Baseline, after four months, and after 12 months, then every year up to 15 years
  Changes in FENO in ppb
Blood Gas Aanalysis | Baseline, four months, yearly for up to 15 years
  pO2 in kPa/ mmHg pCO2 in kPa/ mmHg and Bloodoxygensaturation in %
Leucozytes | Baseline, four months, yearly for up to 15 years
  Changes in Leucozytes in nl
Neutrophilic granulocytes | Baseline, four months, yearly for up to 15 years
  in nl or %
Eosinophilic granulocytes | Baseline, four months, yearly for up to 15 years
  in µl or %
Mortality | Baseline, four months, yearly for up to 15 years
  Mortality rate due to severe Asthma

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Leuppi, Principal Investigator — Kantonsspital Baselland Liestal
Locations (10):
- Switzerland (10):
  - Cantonal Hospital Baselland Liestal, Liestal, Basel-Landschaft
  - Universitätsklinik für Pneumologie, Inselspital, Bern
  - Pneumologie, Kantonsspital Graubünden, Chur
  - Klinik für Pneumologie, Hochgebirgsklinik Davos, Davos
  - Hôpitaux Universitaires Genève, Geneva
  - Centre hospitalier universitaire vaudoise, Lausanne
  - Pneumologia, Ospedale Civico, Lugano
  - Klinik für Pneumologie und Schlafmedizin, Kantonsspital St.Gallen, Sankt Gallen
  - Hôpital du valais, sion, Sion
  - Klinik für Pneumologie, Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided